CLINICAL TRIAL: NCT00724841
Title: A Multi-Center, Open-Label, Phase I/II Study of GEM1777 in Combination With Temozolomide Administered Every 4 Weeks to Patients With Metastatic Melanoma
Brief Title: A Phase I/II Study of GMX1777 in Combination With Temozolomide for the Treatment of Metastatic Melanoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study terminated prematurely due to financial contraints.
Sponsor: Gemin X (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEM303
Record Dates: First submitted 2008-07-28; First posted 2008-07-30 (Estimated); Last update posted 2016-07-22 (Estimated); Status verified 2016-07

CONDITIONS: Metastatic Melanoma
MeSH Terms: conditions — Melanoma | interventions — obatoclax; 1-(2-(2-(2-(2-methoxyethoxy)ethoxy)ethoxy)ethoxycarbonyloxymethyl)-4-(N'-cyano-N''-(6-(4-chlorophenoxy)hexyl)-N-guanidino)pyridinium; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- 1 (Experimental): 40 mg/m2 GMX1777 with Temozolomide
  Interventions: Drug: Obatoclax Mesylate; Drug: Temozolomide
- 2 (Experimental): 50 mg/m2 GMX1777 with Temozolomide
  Interventions: Drug: Obatoclax Mesylate; Drug: Temozolomide
- 3 (Experimental): 62 mg/m2 GMX1777 with Temozolomide
  Interventions: Drug: Obatoclax Mesylate; Drug: Temozolomide
- 4 (Experimental): 80 mg/m2 GMX1777 with Temozolomide
  Interventions: Drug: Obatoclax Mesylate; Drug: Temozolomide
- 5 (Experimental): 100 mg/m2 GMX1777 with Temozolomide
  Interventions: Drug: Obatoclax Mesylate; Drug: Temozolomide
- 6 (Experimental): 125 mg/m2 GMX1777 with Temozolomide
  Interventions: Drug: Obatoclax Mesylate; Drug: Temozolomide

INTERVENTIONS:
Drug: Obatoclax Mesylate — Obatoclax Mesylate (GMX1777) at various doses in combination with temozolomide
  Other Names: GMX1777
Drug: Temozolomide

SUMMARY:
Obatoclax Mesylate (GMX1777) is a water-soluble, intravenously-administered pro-drug of GMX1778. GMX1777 is rapidly converted to GMX1778 in vivo. GMX1778 has potent anti-tumor activity against a variety of cell lines and models from different tumor origins.

DETAILED DESCRIPTION:
GMX1777 will be administered as 3-Hour Infusions in Combination with Temozolomide taken orally for the treatment of Metastatic Melanoma. GMX1777 infusion will be given on either day 1, days 1 and 3, or days 1,3, and 5 every 4 weeks. Temozolomide will be administered on 5 consecutive days every 4 weeks. No investigational or commercial agents or therapies other than those described may be administered with the intent to treat the patient's malignancy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed metastatic melanoma
* Up to 1 prior chemotherapy regimen allowed; prior immunotherapy allowed
* Normal organ and marrow function
* Willing to submit to blood sampling for planned PK/PD analyses
* Ability of understand and willingness to sign a written informed consent

Exclusion Criteria:

* No other investigational or commercial agents or therapies
* Prior exposure to GMX1777, GMX1778 or CHS828
* Patients with uncontrolled, intercurrent illness
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2008-06; Primary Completion 2008-07 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Determine the recommended Phase II dose of GMX1777 in combination with temozolomide | 2 years
Learn more about the side effects of taking GMX1777 in combination with temozolomide | Within the first 4 weeks
Determine the disease response to treatment with GMX1777 in combination with temozolomide | Within the first 8 weeks

SECONDARY OUTCOMES:
Learn more about how the body processes GMX1777 | Within the fisrt 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Mark Berger, MD, Study Director — Gemin X, Inc.
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States